CLINICAL TRIAL: NCT01763203
Title: Secondary Stroke Prevention by Uniting Community and Chronic Care Model Teams Early to End Disparities: the SUCCEED Trial
Brief Title: The SUCCEED Trial of Secondary Stroke Prevention
Acronym: SUCCEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: University of Southern California (Other); Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other); Rancho Los Amigos National Rehabilitation Center (Other); Olive View-UCLA Education & Research Institute (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); California Community Foundation (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Barbara Vickrey, MD, MPH, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5155 U54-NS081764; U54NS081764 (NIH)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Stroke; Secondary Stroke Prevention
Keywords: Self-management; Chronic Care Model; Community health worker
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care Management+Community Health Worker (Experimental): Care management
  Interventions: Behavioral: Care Management+Community Health Worker
- Usual Care (Active Comparator): Written materials
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Care Management+Community Health Worker — Over a period of a year subjects randomized into the Intervention arm of the study will receive support from a Care Manager. Subjects will also participate in educational group sessions on chronic disease self-management and have home visits by a Community Health Worker who will use mobile health technology.
  Arms: Care Management+Community Health Worker
Behavioral: Usual Care — Subjects randomized into the Usual Care arm will receive educational materials about stroke distributed to the Intervention patients and will receive their post-stroke care as usual.
  Arms: Usual Care

SUMMARY:
The purpose of this study is to test a newly-developed outpatient clinic and community-based care intervention called SUCCEED (Secondary stroke prevention by Uniting Community and Chronic care model teams Early to End Disparities) for improving control of stroke risk factors among stroke patients in the Los Angeles County "safety net", and to measure the costs of running such an intervention, relative to usual care.

DETAILED DESCRIPTION:
Individuals randomized to the intervention arm will receive care from a team that consists of a care manager(CM) who is either a nurse practitioner (NP) or physician assistant (PA), supervised by the site PI, and a community health worker (CHW). The CM will follow care protocols developed by the research team. The CHW will serve as a liaison between the patient and the health care system, and mobilize resources and system support to reduce social isolation and improve stroke risk factor control self-management, through a series of workshops and home visits. Intervention participants will receive home blood pressure monitors. Subjects in either arm are eligible to receive their usual source of care. Five hundred participants who have had a stroke or TIA will be enrolled, randomized to the intervention or to usual care in a 1:1 ratio, and followed for 12 months. The impact of the intervention on systolic blood pressure is the primary study outcome; secondary outcomes are other stroke risk factors. Enrollment will occur at four sites in Los Angeles County, and the study sample is projected to include over 90% socioeconomically disadvantaged individuals from minority groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Los Angeles County+University of Southern California (LAC-USC), Rancho Los Amigos, Olive View-University of California, Los Angeles (UCLA), or Harbor-UCLA
* Transient ischemic attack (TIA), ischemic stroke or hemorrhagic stroke within the prior 90 days
* English, Spanish, Korean, Mandarin or Cantonese-speaking
* 40 years of age or older
* Capable of giving informed consent (no proxies will be used to obtain consent)
* Systolic blood pressure is 130 mm Hg or greater OR Systolic blood pressure is between 120 mm Hg and 130 mm Hg and there is diagnosed/treated hypertension prior to the stroke or TIA

Exclusion Criteria:

* Younger than 40 years
* Systolic Blood Pressure less than 120 mm Hg OR systolic blood pressure is between 120 mm Hg and 130 mm Hg and there is no known history of hypertension prior to the stroke or TIA
* Speaks language other than English, Spanish, Korean, Mandarin, and Cantonese
* Inability to comprehend the study because of communication or cognitive impairments

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2014-02-13 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara G Vickrey, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Amytis Towfighi, MD, Principal Investigator — USC - Department of Neurology. Rancho Los Amigos National Rehabilitation Center
Locations (6):
- United States (6):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - UCLA, Los Angeles, California
  - LAC+USC Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Olive View-UCLA Medical Center, Sylmar, California
  - Harbor-UCLA Medical Center, Torrance, California

REFERENCES:
- [Background] Towfighi A, Cheng EM, Ayala-Rivera M, McCreath H, Sanossian N, Dutta T, Mehta B, Bryg R, Rao N, Song S, Razmara A, Ramirez M, Sivers-Teixeira T, Tran J, Mojarro-Huang E, Montoya A, Corrales M, Martinez B, Willis P, Macias M, Ibrahim N, Wu S, Wacksman J, Haber H, Richards A, Barry F, Hill V, Mittman B, Cunningham W, Liu H, Ganz DA, Factor D, Vickrey BG. Randomized controlled trial of a coordinated care intervention to improve risk factor control after stroke or transient ischemic attack in the safety net: Secondary stroke prevention by Uniting Community and Chronic care model teams Early to End Disparities (SUCCEED). BMC Neurol. 2017 Feb 6;17(1):24. doi: 10.1186/s12883-017-0792-7. PMID 28166784
- [Background] Schneider AT, Pancioli AM, Khoury JC, Rademacher E, Tuchfarber A, Miller R, Woo D, Kissela B, Broderick JP. Trends in community knowledge of the warning signs and risk factors for stroke. JAMA. 2003 Jan 15;289(3):343-6. doi: 10.1001/jama.289.3.343. PMID 12525235
- [Background] Lu M, Safren SA, Skolnik PR, Rogers WH, Coady W, Hardy H, Wilson IB. Optimal recall period and response task for self-reported HIV medication adherence. AIDS Behav. 2008 Jan;12(1):86-94. doi: 10.1007/s10461-007-9261-4. Epub 2007 Jun 19. PMID 17577653
- [Background] Simoni JM, Kurth AE, Pearson CR, Pantalone DW, Merrill JO, Frick PA. Self-report measures of antiretroviral therapy adherence: A review with recommendations for HIV research and clinical management. AIDS Behav. 2006 May;10(3):227-45. doi: 10.1007/s10461-006-9078-6. PMID 16783535
- [Background] Nicol MB, Thrift AG. Knowledge of risk factors and warning signs of stroke. Vasc Health Risk Manag. 2005;1(2):137-47. doi: 10.2147/vhrm.1.2.137.64085. PMID 17315400
- [Derived] Saunders DH, Mead GE, Fitzsimons C, Kelly P, van Wijck F, Verschuren O, Backx K, English C. Interventions for reducing sedentary behaviour in people with stroke. Cochrane Database Syst Rev. 2021 Jun 29;6(6):CD012996. doi: 10.1002/14651858.CD012996.pub2. PMID 34184251
- [Derived] Towfighi A, Cheng EM, Ayala-Rivera M, Barry F, McCreath H, Ganz DA, Lee ML, Sanossian N, Mehta B, Dutta T, Razmara A, Bryg R, Song SS, Willis P, Wu S, Ramirez M, Richards A, Jackson N, Wacksman J, Mittman B, Tran J, Johnson RR, Ediss C, Sivers-Teixeira T, Shaby B, Montoya AL, Corrales M, Mojarro-Huang E, Castro M, Gomez P, Munoz C, Garcia D, Moreno L, Fernandez M, Lopez E, Valdez S, Haber HR, Hill VA, Rao NM, Martinez B, Hudson L, Valle NP, Vickrey BG; Secondary Stroke Prevention by Uniting Community and Chronic Care Model Teams Early to End Disparities (SUCCEED) Investigators. Effect of a Coordinated Community and Chronic Care Model Team Intervention vs Usual Care on Systolic Blood Pressure in Patients With Stroke or Transient Ischemic Attack: The SUCCEED Randomized Clinical Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2036227. doi: 10.1001/jamanetworkopen.2020.36227. PMID 33587132
- [Derived] Lin AM, Vickrey BG, Barry F, Lee ML, Ayala-Rivera M, Cheng E, Montoya AV, Mojarro-Huang E, Gomez P, Castro M, Corrales M, Sivers-Teixeira T, Tran JL, Johnson R, Ediss C, Shaby B, Willis P, Sanossian N, Mehta B, Dutta T, Razmara A, Bryg R, Song S, Towfighi A. Factors Associated With Participation in the Chronic Disease Self-Management Program: Findings From the SUCCEED Trial. Stroke. 2020 Oct;51(10):2910-2917. doi: 10.1161/STROKEAHA.119.028022. Epub 2020 Sep 11. PMID 32912091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The dates of the recruitment period are from February 13, 2014 through August 31, 2017.
Pre-assignment Details: Not applicable; all enrolled participants were assigned to an arm.
Period: Overall Study
Arm/Group | Care Management+Community Health Worker | Usual Care
Started | 241 | 246
Completed | 208 | 204
Not Completed | 33 | 42
Not completed — Death | 4 | 7
Not completed — Lost to Follow-up | 12 | 12
Not completed — Withdrawal by Subject | 8 | 12
Not completed — Moved out of study region | 7 | 10
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Population: Not applicable - analysis population is different from participants enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Care Management+Community Health Worker | Usual Care | Total
Number analyzed (Participants) | 241 | 246 | 487
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (9.0) | 57.0 (8.7) | 57.1 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 92 | 170
  Male | 163 | 154 | 317
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 170 | 177 | 347
  Not Hispanic or Latino | 71 | 69 | 140
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 15 | 15 | 30
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 5
  Black or African American | 45 | 42 | 87
  White | 168 | 167 | 335
  More than one race | 3 | 7 | 10
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 241 | 246 | 487
Index vascular event [Count of Participants; unit: Participants]
  Ischemic stroke | 190 | 193 | 383
  Intracerebral hemorrhage | 40 | 38 | 78
  Transient ischemic attack | 11 | 15 | 26
Survey language [Count of Participants; unit: Participants]
  English | 101 | 106 | 207
  Spanish | 140 | 140 | 280
Location of birth [Count of Participants; unit: Participants]
  Born in the US | 65 | 69 | 134
  Born outside of the US | 176 | 176 | 352
  Not reported | 0 | 1 | 1
Employment status prior to vascular event [Count of Participants; unit: Participants]
  Working for pay | 125 | 141 | 266
  Not working for pay | 115 | 102 | 217
  Not reported | 1 | 3 | 4
Education [Count of Participants; unit: Participants]
  Bachelor's degree and higher | 33 | 22 | 55
  Some college | 29 | 37 | 66
  High school graduate/GED (no college) | 15 | 22 | 37
  Some high school but not a high school graduate | 59 | 56 | 115
  First to eighth grade | 78 | 82 | 160
  No school/kindergarten only | 12 | 11 | 23
  Not reported | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Systolic Blood Pressure
Description: Blood pressure at 12 months will be the primary outcome. Blood pressure will also be measured at baseline and at the 3-month mark to track blood pressure during the entire participation period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
mm Hg | 133.1 (20.5) | 136.9 (21.9)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.73, Mixed Models Analysis

2. Secondary Outcome: Dyslipidemia
Description: non-HDL cholesterol will be measured at 12-months. The same measurements will be taken at baseline and at the 3 month mark in order to track measurements throughout the entire participation period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
mg/dL | 98.7 (47.8) | 104.1 (49.2)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.77, Mixed Models Analysis

3. Secondary Outcome: Percentage of Glycated Hemoglobin (Hemoglobin A1C)
Description: Hemoglobin A1C will be measured at 12-months. The same measurements will be taken at baseline and at the 3 month mark in order to track measurements throughout the entire participation period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: percentage of glycated hemoglobin
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
percentage of glycated hemoglobin | 6.5 (1.2) | 6.6 (1.3)

4. Secondary Outcome: Inflammation: C-reactive Protein
Description: C-reactive protein will be measured at 12-months. The same measurements will be taken at baseline and at the 3 month mark in order to track measurements throughout the entire participation period.
Time Frame: 12 months
Measure: Geometric Mean (Standard Deviation); unit: mg/L
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
mg/L | 1.1 (3.2) | 1.2 (3.2)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.002, Mixed Models Analysis

5. Secondary Outcome: Body Mass Index
Description: Body mass index will be measured at 12-months with a height and weight ratio. The same measurements will be taken at baseline and at the 3 month mark in order to track measurements throughout the entire participation period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg/meter^2
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
kg/meter^2 | 29.5 (5.9) | 29.2 (5.1)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.86, Mixed Models Analysis

6. Secondary Outcome: Waist Circumference
Description: Waist circumference will be measured at 12-months according to the National Institutes of Health (NIH) guidelines. The same measurements will be taken at baseline and at the 3 month mark in order to track measurements throughout the entire participation period.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
cm | 102.9 (14.3) | 101.4 (12.5)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.10, Mixed Models Analysis

7. Secondary Outcome: Physical Activity
Description: The International Physical Activity Questionnaire (IPAQ) Short 7-Day version will be collected as part of the 12 month outcome survey. The questionnaire will also be collected at baseline and 3 months to track changes over the entire study period. The IPAQ score reflects energy expenditure of physical activity, and is reported in units of 'met minutes' which means metabolic equivalent. The minimum value is zero and there is no maximum. Higher scores mean better levels of physical activity.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: IPAQ met minutes
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
IPAQ met minutes | 1251 (1808) | 1344 (1874)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.46, Mixed Models Analysis

8. Secondary Outcome: Salt Intake
Description: A single question, "Are you currently watching or reducing your sodium or salt intake?" from the Behavioral Risk Factor Surveillance System 2013, which has a dichotomous 'yes/no' response, will be collected as part of the 12 month outcome survey. The question will also be collected at baseline, 3 months, and at 8 months, to track changes over the entire study period
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  Yes | 181 | 168
  No | 27 | 34
  unknown | 33 | 44
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.011, Mixed Models Analysis

9. Secondary Outcome: Soda Intake
Description: A single question from the California Health Interview Survey (CHIS) 2011-2012 will be collected as part of the 12-month outcome survey. The question is "During the past month, how often did you drink regular soda or pop that contains sugar?" The participant gives a number, and the frequency (per day, per week, or per month) is also recorded. The average daily servings of soda over the prior month is calculated, and the question is scored as a dichotomous variable of greater than or equal to 1 serving of soda per /day versus less than one serving of soda per day. The question will also be collected at baseline and at 3 months, to track changes over the entire study period
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  No soda servings per day in past month | 107 | 102
  Any soda servings per day over past month | 99 | 99
  Unknown | 35 | 45
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.47, Mixed Models Analysis

10. Secondary Outcome: Fruit and Vegetable Intake
Description: Two questions from the California Health Interview Survey (CHIS) 2011-2012 will be collected as part of the 12-month outcome survey. The questions are "During the past month, how many times did you eat fruit? Do not count juices" and "During the past month, how many times did you eat any other vegetables like green salad, green beans or potatoes? Do not include fried potatoes." For each question, the participant gives a number, and the frequency (per day, per week, or per month) is also recorded. Responses are converted to a number for day for each question, then summed across the two questions. The question is scored as a dichotomous variable of five or more servings of fruit and vegetables per day versus less than five servings of fruit and vegetables per day. The questions will also be collected at baseline and at 3 months, to track changes over the entire study period
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  >= 5 fruit+vegetables servings/day in past month | 22 | 28
  <5 fruit+vegetables servings/day in past month | 184 | 172
  unknown | 35 | 46
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.58, Mixed Models Analysis

11. Secondary Outcome: Smoking
Description: A single question from the California Health Interview Survey 2011-2012 Adult Questionnaire will be collected as part of the 12-month outcome survey. The question asks whether over the interval since the previous study interview, "were you smoking cigarettes every day, some days, or not at all?" The question will also be collected at baseline (with a time frame of over the prior year) and at 3 months, to track changes over the entire study period. The scoring for this outcome is dichotomous: "Smoking" = a response of 'every day' or 'some days', versus "Not smoking" = a response of 'not at all.'
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  Smoking | 25 | 22
  Not smoking | 182 | 181
  Unknown | 34 | 43
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.74, Mixed Models Analysis

12. Secondary Outcome: Knowledge About Stroke Signs
Description: An open-ended question about what the participant believes is a sign of a stroke ("What are the warning signs of a stroke? What else...what else?"), will be asked as a part of the 12 month survey. This question will also be collected at 3 months to track changes over the follow-up study period. Correct responses are numbness, weakness, difficulty speaking/understanding, vision disturbance, dizziness, and headache. Responses are scored as 0 correct, 1 correct, 2 correct, and 3 or more correct.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  3 or more correct stroke signs | 95 | 65
  2 correct stroke signs | 69 | 75
  1 correct stroke sign | 28 | 40
  no correct stroke sign | 16 | 24
  unknown | 33 | 42
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.0021, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Knowledge About Stroke Risk Factors
Description: An adaptation of an existing instrument will be collected as a part of the 12 month survey. An open-ended question about what the participant believes is a stroke risk factor ("I would like to ask you about stroke risk factors, those are the things that make it more likely for somebody to have a stroke. From anything you might have heard or read, what do you believe are the risk factors associated with stroke? What else...what else?", will be asked, then converted to three dichotomous variables: correct about at least 3 stroke risk factors versus less than three; correct about at least one stroke risk factor versus none correct; and reports that blood pressure is a stroke risk factor versus does not. This question will also be collected at baseline, 3 months, and 8 months to track changes over the entire study period.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  at least 3 correct stroke risk factors named | 54 | 49
  less than 3 correct stroke risk factors named | 154 | 155
  unknown | 33 | 42
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.07, Mixed Models Analysis

14. Secondary Outcome: Patient Perception of Quality of Stroke Preventative Care
Description: An adaptation of the Consumer Assessment of Healthcare Providers and Systems (CAHPS) will be collected as a part of the 12 month questionnaire. It will also be collected at baseline and 3 month to track changes over the entire study period. The CAHPS question was "Did you receive from any of your medical care providers the help you needed to make changes in your habits or lifestyle that would improve your health or prevent illness?" Response choices are: 'Yes definitely' "Yes somewhat' or 'No definitely not'.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  Yes, definitely | 126 | 91
  Yes, somewhat | 30 | 42
  No, definitely not | 36 | 55
  Unknown | 49 | 58
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.32, Mixed Models Analysis

15. Secondary Outcome: Vascular Events
Description: The Questionnaire for Verifying Stroke Free Status (QVSFS) will be collected as part of the 12 month survey. It will also be collected at baseline and 3 months to track changes over the entire study period. This questionnaire will also be collected every 6 months for up to 24 months after the study is completed to check for vascular events. The scoring was dichotomous: at least one new event (stroke, transient ischemic attack, or heart attack) versus none over the 12-month follow-up period.
Time Frame: 12 months
Population: This outcome was only assessed during follow-up, so participants with no follow-up data (ie only baseline data) were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 220 | 225
Participants
  >=one vascular event during the 12-month follow-up | 26 | 29
  No vascular events during the 12-month follow-up | 194 | 196
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.77, Chi-squared

16. Secondary Outcome: Medication Adherence - Global
Description: A single item adapted from two questions published elsewhere will be administered at 12 months. The adapted item is "In the past week, how much of the time were you able to take your medications exactly as your doctor or nurse told you to?" Response choices are 'None of the time,' 'A little of the time,' "A good bit of the time,' 'Most of the time,' or 'All of the time.' This item will also be collected at Baseline, 3 Months, and 8 Months, to track changes over the entire study period.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 241 | 246
Participants
  All of the time | 148 | 150
  Most of the time | 31 | 27
  A good bit of the time | 2 | 1
  A little of the time | 7 | 9
  None of the time | 7 | 4
  Unknown | 46 | 55
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.20, Mixed Models Analysis

17. Secondary Outcome: Medication Adherence - Blood Pressure Medication
Description: A continuous measure of adherence as percentage of doses taken over the prior 7-day time period will be collected at 12 months and calculated for blood pressure medication, using a previously published formula. This will also be collected at 3 months, to track changes over the study period.
Time Frame: 12 Months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 161 | 161
percentage of doses | 91.6 (24) | 89.4 (27)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.45, t-test, 2 sided

18. Secondary Outcome: Medication Adherence - Cholesterol Medication
Description: A continuous measure of adherence as percentage of doses taken over the prior 7-day time period will be collected at 12 months and calculated for cholesterol medication, using a previously published formula. This will also be collected at 3 Months, to track changes over the study period.
Time Frame: 12 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 153 | 146
percentage of doses | 86.7 (32) | 87.1 (32)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.93, t-test, 2 sided

19. Secondary Outcome: Medication Adherence - Antithrombotic Medication
Description: A continuous measure of adherence as percentage of doses taken over the prior 7-day time period will be collected at 12 months and calculated for antithrombotic medication, using a previously published formula. This will also be collected at 3 Months, to track changes over the study period.
Time Frame: 12 months
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 152 | 153
percentage of doses | 88.5 (30) | 89.4 (29)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.80, t-test, 2 sided

20. Secondary Outcome: Medication Adherence - Antidepressant Medication
Description: A continuous measure of adherence as percentage of doses taken over the prior 7-day time period will be collected at 12 months and calculated for antidepressant medication, using a previously published formula. This will also be collected at 3 Months, to track changes over the study period.
Time Frame: 12 months
Population: Only study participants taking antidepressant medication were included in this analysis
Measure: Mean (Standard Deviation); unit: percentage of doses
Arm/Group | Care Management+Community Health Worker | Usual Care
Number analyzed (Participants) | 28 | 25
percentage of doses | 87.8 (32) | 96.2 (20)
Statistical Analysis 1: Comparison: Care Management+Community Health Worker vs Usual Care; Test type: Superiority; p = 0.25, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Care Management+Community Health Worker | Usual Care
All-Cause Mortality (participants affected / at risk) | 4/241 | 7/246
Serious Adverse Events (participants affected / at risk) | 0/241 | 0/246
Other Adverse Events (participants affected / at risk) | 0/241 | 0/246

LIMITATIONS AND CAVEATS:
The primary study limitation was the lack of full implementation of the multi-component care management interventions within the intervention arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT01763203/Prot_SAP_000.pdf